CLINICAL TRIAL: NCT05953311
Title: The Relationship Between Neurological Blood-based Biomarkers and Mid-term Cognitive Disorders in Critically Ill Survivors.
Brief Title: Neurological Blood-based Biomarkers and Cognitive Disorders in Critically Ill Survivors.
Acronym: COGNISI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Sponsor
Other Study IDs: COGNISI
Record Dates: First submitted 2023-06-29; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Intensive Care Unit Syndrome; Post-intensive Care Syndrome; Cognitive Disorder
MeSH Terms: conditions — postintensive care syndrome; Cognitive Dysfunction | interventions — Hematologic Tests; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU survivors: Cohort of patients who survive an ICU stay of at least 7 days
  Interventions: Other: Blood analysis; Other: Cognitive tests

INTERVENTIONS:
Other: Blood analysis — Blood analysis for neurological biomarkers measurements
Other: Cognitive tests — Questionnaires assessing cognitive function

SUMMARY:
Cognitive disorders are common after intensive care. Currently, their diagnosis is based on clinical tests. The investigators plan to study the relationship between different neurological blood biomarkers (cytokines, S100β protein, neuron specific enolase, total Tau protein and neurofilament light chain) and the occurrence of cognitive disorders during the three months following intensive care discharge.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated ICU stay of at least 7 days for sepsis, acute respiratory distress syndrome, severe burns
* French speaking

Exclusion Criteria:

* hearing loss or blindness
* mental retardation
* known cognitive disorders or dementia
* ICU admission for neurological disease
* refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who survive an ICU stay of at least 7 days and who are assessed 3 months after ICU discharge
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood neurological biomarkers levels | ICU Admission
  Measurement of blood levels of S100β protein
Blood neurological biomarkers levels | day 3 after ICU admission
  Measurement of blood levels of S100β protein
Blood neurological biomarkers levels | day 7 after ICU admission
  Measurement of blood levels of S100β protein
Blood neurological biomarkers levels | day 14 after ICU admission
  Measurement of blood levels of S100β protein
Blood neurological biomarkers levels | 3 months after ICU discharge
  Measurement of blood levels of S100β protein
Blood neurological biomarkers levels | ICU Admission
  Measurement of blood levels of neuron specific enolase
Blood neurological biomarkers levels | day 3 after ICU admission
  Measurement of blood levels of neuron specific enolase
Blood neurological biomarkers levels | day 7 after ICU admission
  Measurement of blood levels of neuron specific enolase
Blood neurological biomarkers levels | day 14 after ICU admission
  Measurement of blood levels of neuron specific enolase
Blood neurological biomarkers levels | 3 months after ICU discharge
  Measurement of blood levels of neuron specific enolase
Blood neurological biomarkers levels | ICU Admission
  Measurement of blood levels of total Tau protein
Blood neurological biomarkers levels | day 3 after ICU admission
  Measurement of blood levels of total Tau protein
Blood neurological biomarkers levels | day 7 after ICU admission
  Measurement of blood levels of total Tau protein
Blood neurological biomarkers levels | day 14 after ICU admission
  Measurement of blood levels of total Tau protein
Blood neurological biomarkers levels | 3 months after ICU discharge
  Measurement of blood levels of total Tau protein
Blood neurological biomarkers levels | ICU Admission
  Measurement of blood levels of neurofilament light chain
Blood neurological biomarkers levels | day 3 after ICU admission
  Measurement of blood levels of neurofilament light chain
Blood neurological biomarkers levels | day 7 after ICU admission
  Measurement of blood levels of neurofilament light chain
Blood neurological biomarkers levels | day 14 after ICU admission
  Measurement of blood levels of neurofilament light chain
Blood neurological biomarkers levels | 3 months after ICU discharge
  Measurement of blood levels of neurofilament light chain
Cognitive disorders assessment (global assessment) | the day after ICU discharge
  Administration of the MOCA questionnaire (Montreal Cognitive Assessment) : scoring from 0 to 30, the highest score meaning the better cognitive outcome)
Cognitive disorders assessment (global assessment) | 3 months after ICU discharge
  Administration of the MOCA questionnaire (Montreal Cognitive Assessment) : scoring from 0 to 30, the highest score meaning the better cognitive outcome)
Memory disorder assessment | 3 months after ICU discharge
  Administration of the California Verbal Learning Test: a Z-score will be used to score this item
Memory disorder assessment | 3 months after ICU discharge
  Administration of the Brief Visuospatial Memory Test (a Z-score will be used to score this item)
Speed of information processing assessment | 3 months after ICU discharge
  Administration of the Ways IV test (a Z-score will be used to score this item)
Executive function assessment | 3 months after ICU discharge
  Administration of the Trail Making Test (a Z-score will be used to score this item)
Memory disorder assessment | 3 months after ICU discharge
  Administration of the Reading Span (working memory) test (a Z-score will be used to score this item)
Executive function assessment | 3 months after ICU discharge
  Administration of the Stroop Color and Word Test (a Z-score will be used to score this item)
Executive function assessment | 3 months after ICU discharge
  Administration of the Go/No-go test (a Z-score will be used to score this item)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Rousseau, MD, PhD, Study Director — University hospital of Liège
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No